CLINICAL TRIAL: NCT03133585
Title: Non-Interventional, International, Post-Marketing Clinical Follow-up Study on the Stoma Appliance Flexima®/Softima® 3S
Brief Title: Study on the Stoma Appliance Flexima®/Softima® 3S
Acronym: KISSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BBraun Medical SAS (Industry)
Collaborators: VERTICAL (Unknown); EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: OPM-O-H-1502
Record Dates: First submitted 2017-04-07; First posted 2017-04-28 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Ostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 2 piece appliance for stomy — Use of the Flexima®/Softima® 3S during 6 months following the patient's usually frequency of appliance change

SUMMARY:
To evaluate the satisfaction of patients of the Flexima®/Softima® 3S with 6 months follow-up.

The primary variable is to evaluate the degree of satisfaction of patients in terms of leakage prevention, comfort and patient's feeling of security to the Flexima®/Softima® 3S.

DETAILED DESCRIPTION:
The primary variable is to evaluate the degree of satisfaction of patients in terms of leakage prevention, comfort and patient's feeling of security to the Flexima®/Softima® 3S.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old
* Patient who has had a colostomy or an ileostomy or a jejunostomy or an urostomy for at least 1 month
* Patient agreeing to participate to the study and having signed the informed consent form/information letter in accordance with local requirements
* Patient for whom the use of Flexima®/Softima® 3S has already been decided within the regular planning of his treatment

Exclusion Criteria:

* Patient with cognitive problems, according to the investigator, preventing him from answering a questionnaire or for whom the evaluation could be a problem
* Patient taking part in another clinical evaluation
* Patient having more than one stomy
* Patient vulnerable and under legal protection
* Patient having had an known allergy to one of the components of the appliance
* Patient previously using Flexima®/Softima® 3S

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a Enterostomy or an urostomy
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2017-08-23 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
evaluation of the satisfaction of patients of the Flexima®/Softima® 3S with 6 months follow-up | the questions will be asked to the patient at each follow up visits (= at 1 month, 3 months and 6 months).Total Score will range from 3 to 12. A total score of 9 or more will define appropriate overall satisfaction.
  The primary variable is to evaluate the degree of satisfaction of patients in terms of leakage prevention, comfort and patient's feeling of security to the Flexima®/Softima® 3S. For each item, the patient will evaluated the product thanks to a 4 points scale question (very good (4)/good(3)/ poor(2)/ very poor(1))

CONTACTS AND LOCATIONS:
Overall Officials: Danièle Chaumier, Principal Investigator — Hopital Tenon, Paris, France
Locations (2):
- France (2):
  - CHU Lapeyronie, Montpellier
  - Hopital Tenon, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No